CLINICAL TRIAL: NCT05541445
Title: A Prospective, Single-arm Phase Ib/II Study to Explore the Safety and Efficacy of Pembrolizumab Combined With Neoadjuvant Chemoradiotherapy (CRT) Followed by Surgery for Upper Locally Advanced Esophageal Squamous Cell Carcinoma (ESCC)
Brief Title: Pembrolizumab Plus CRT Followed by Surgery in Upper ESCC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Upper EC program
Record Dates: First submitted 2022-09-13; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Immunotherapy combined with chemotherapy and radiotherapy
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — The subjects first receive induction therapy with pembrolizumab combined with chemotherapy for 6 weeks, and then receive sequential therapy with pembrolizumab combined with concurrent chemoradiotherapy for 6 weeks, and receive surgical treatment within 4-8 weeks after neoadjuvant therapy. For patients whose postoperative pathology is confirmed as PCR (pathological complete response), the patients will be observed with long-time follow-up; If the postoperative pathology is confirmed as non-PCR, pembrolizumab will be administrated until 1 year or disease progression or intolerable toxicity.
  Other Names: IO combined therapy

SUMMARY:
Through a prospective, single-center, single-arm, phase Ib/II study, we aim to explore the safety and feasibility of a new treatment mode for upper esophageal cancer, which is that pembrolizumab combined with chemoradiotherapy as neoadjuvant therapy and then followed by radical surgery.

DETAILED DESCRIPTION:
Treatment includes induction treatment, sequential treatment and maintenance treatment.

1. Preoperative neoadjuvant therapy 1) Induction therapy (2 cycles): Immunotherapy+Chemotherapy Pembrolizumab 200mg, IV, D1, q3w, Albumin paclitaxel, 125mg/m2, IV, D1/D8, q3w; Cisplatin, 70mg/m2 in total, IV, given in three times, q3w. 2) Sequential treatment: Immunotherapy+Chemoradiotherapy Pembrolizumab 200mg, IV, D1, q3w, 2 cycles; Albumin paclitaxel, 100mg, IV, D1, QW, 4 cycles; Cisplatin, 20mg/m2, IV, D1, QW, 4 cycles. Radiotherapy: PTV: 44gy/2gy/22fx, 5 days a week, 5 weeks in total.
2. Surgery 4-8 weeks after the end of the neoadjuvant therapy, the operation can be performed only when the indexes of leukocyte, platelet, liver and kidney function of the patient are normal. The operation aims to achieve R0 resection with laryngeal preservation.
3. Postoperative adjuvant treatment Patients who did not reach pCR after operation were given pembrolizumab 200mg, IV, D1, q3w 4-6 weeks after operation until 1 year, disease progression or intolerable toxicity.
4. Follow-up period Patients will be continuously monitored during the study. The enrolled subjects will be closely followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before enrollment;
2. Be aged 18-80 years old, and be male or female;
3. Have potentially upper ESCC (upper edge of tumor ≤ 5cm from esophageal entrance) diagnosed with cT1-3N1-2M0 or cT2-3N0M0 (AJCC 8th);
4. Have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-1;
5. No previous treatments;
6. Be eligible for R0 resection before treatment;
7. Demonstrate adequate organ function; all screening laboratory tests will be performed within 10 days of treatment initiation;
8. Have a negative urine or serum pregnancy within 72 hours before receiving the first dose of study medication if they are a female subject with childbearing potential. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required;
9. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion through repeated biopsies. "Newly obtained" is defined as a specimen obtained up to 4 weeks (28 days) before the initiation of treatment on Day 10. Subjects for whom newly obtained samples cannot be provided (e.g., as newly obtained sample is inaccessible or due to subject safety concerns) may submit an archived specimen, but only with the agreement of the sponsor;

11. Be expected to survive >6 months; 12. Join the clinical study on a completely voluntary basis, demonstrate good adherence, and cooperate with the follow-up assessments for safety and survival

Exclusion Criteria:

1. Have undergone any previous therapy (e.g., an operation, radiotherapy, immunotherapy, or chemotherapy) for ESCC;
2. Have a history of other malignant tumor;
3. Be ineligible or have a contraindication for esophagectomy;
4. Have a history of other anti-PD-1/PD-L1 therapies, or have a known history of an allergy to macromolecular protein preparations or any component of PD-1;
5. Have a diagnosis of immunodeficiency or have received chronic systemic steroid therapy (in doses >10 mg daily of a prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of the study drug;
6. Have an active autoimmune disease that required systemic treatment in the past 2 years (e.g., the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs);
7. Have poorly controlled cardiac symptoms or cardiac diseases;
8. Have a history or evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, or severely impaired lung function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | 4 months
  Viable tumor comprised ≤ 10% of resected tumor specimens

SECONDARY OUTCOMES:
R0 resection rate | At time of surgery
  R0 resection rate
Larynx preservation rate | At time of surgery
  Larynx preservation rate
Disease-free survival (DFS) | 24 months
  DFS is defined as the time interval between the date of enrollment and the date of the first documented evidence of relapse after radical resection at any site or death related to cancer (including toxicity), whichever occurred first.
Local-regional recurrence free survival (LRRFS) | 24 months
  LRRFS is defined as the time interval between the date of enrollment and the date of the first documented evidence of local-regional relapse after radical resection at primary site or death related to cancer (including toxicity), whichever occurred first.
Overall survival (OS) | 24 months
  Time from the enrollment to death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jie He, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No